CLINICAL TRIAL: NCT00460174
Title: A Phase II Trial of Weekly Gemcitabine Hydrochloride and Bevacizumab in Combination With Abdominal Radiation Therapy in Patients With Localized Pancreatic Cancer
Brief Title: Gemcitabine, Bevacizumab, and Abdominal Radiation Therapy in Treating Patients With Localized Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 04I6; NU-04I6; STU00006774 (Other: Northwestern University IRB)
Record Dates: First submitted 2007-04-11; First posted 2007-04-13 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Pancreatic Cancer
Keywords: stage I pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Bevacizumab; Gemcitabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental): Concurrent gemcitabine, bevacizumab, and radiation therapy
  Interventions: Biological: bevacizumab; Drug: gemcitabine; Procedure: conventional surgery; Radiation: radiation therapy

INTERVENTIONS:
Biological: bevacizumab — 10 mg/kg every 2 weeks as an intravenous infusion after gemcitabine and before radiation
  Other Names: Avastin
Drug: gemcitabine — 1000 mg/m2, 30 minute intravenous infusion, cycle 1 (weeks 1, 2), cycle 2 (weeks 4, 5, 6) and cycle 3 (weeks 8 and 9). During cycle 2, gemcitabine will be delivered prior to radiation therapy
  Other Names: gemcitabine hydrochloride
Procedure: conventional surgery — If resectable, patients will undergo surgery no less than 6 weeks following last dose of bevacizumab. Unresectable patients will not undergo surgery.
Radiation: radiation therapy — 2.4 Gy fractions, 5 fractions/week during cycle 2 only (weeks 4, 5, 6). Total dose 36 Gy.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the tumor growth by blocking blood flow to the tumor. Radiation therapy uses high-energy x-rays to kill tumor cells. Gemcitabine and bevacizumab may make tumor cells more sensitive to radiation therapy. Giving gemcitabine together with bevacizumab and radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving gemcitabine together with bevacizumab and abdominal radiation therapy works in treating patients with localized pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the objective response rate in patients treated with concurrent bevacizumab, gemcitabine hydrochloride, and abdominal radiotherapy.

Secondary

* Determine the quantitative toxicity associated with the delivery of this regimen in these patients.
* Determine the 1-year and median survival of patients treated with this regimen.
* Determine the time to progression in patients treated with this regimen.
* Determine the patterns of recurrence in the entire population of patients treated with this regimen and in the subgroup that is resected for cure.
* Determine the safety of this regimen in these patients.
* Evaluate the surgical experience of patients who undergo surgical resection after completion of protocol-directed therapy.
* Evaluate the toxicity associated with surgical resection in these patients.

OUTLINE: Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 of courses 1 and 3 and on days 1, 8, and 15 of course 2. Patients also receive bevacizumab IV over 30-90 minutes on days 1 and 15 of course 1, on days 8 and 22 of course 2, and on day 8 of course 3. Treatment repeats every 3-4 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity. Beginning on day 1 of the second course of chemotherapy, patients undergo concurrent abdominal radiotherapy once daily, five days a week, for 3 weeks.

Patients are evaluated at week 10. Patients whose disease deemed resectable after study treatment undergo standard pancreatic resection at least 6 weeks after completion of bevacizumab. Patients who remain unresectable and have not progressed after completion of chemoradiotherapy may begin maintenance therapy comprising gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15 and bevacizumab IV over 30-90 minutes on days 1 and 15. Treatment with gemcitabine hydrochloride and bevacizumab repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed periodically for up to 10 years.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of localized pancreatic cancer

  * No metastatic disease
* Resectable or unresectable tumor based on spiral CT with both oral and intravenous contrast enhancement, defined by the following National Comprehensive Cancer Network (NCCN) criteria for resectability*:

  * Resectable tumors meeting the following criteria:

    * No distant metastases
    * Clear fat plane around celiac and superior mesenteric arteries
    * Patent superior mesenteric vein/portal vein
  * Tumors considered borderline resectable according to NCCN criteria, including any of the following, are considered unresectable for the purpose of this study:

    * Severe unilateral superior mesenteric vein/portal impingement
    * Tumor abutment on the superior mesenteric artery
    * Gastroduodenal artery encasement up to the origin at the hepatic artery
    * Colon invasion NOTE: *Determination of resectability must be made prior to study entry based on NCCN criteria
* Patients with biliary or gastroduodenal obstruction must have drainage or surgical bypass prior to starting chemoradiotherapy
* Radiographically assessable disease

  * Malignant disease must be encompassable within a single irradiation field
* No gross duodenal invasion noted on endoscopy
* No CNS or brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for up to 3 months after completion of study therapy
* Bilirubin ≤ 2.0 mg/dL
* AST or ALT ≤ 2.5 times upper limit of normal
* Urine protein:creatinine ratio < 1.0
* Proteinuria < 2+ by dipstick urinalysis OR baseline protein ≤ 1 g/24-hour urine collection
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9.0 g/dL (transfusion or epoetin alfa support allowed)
* INR ≤ 1.5
* No other malignancy within the past 5 years except nonmelanomatous skin cancer or carcinoma in situ of the cervix, uterus, or bladder
* No concurrent significant infection or other medical condition that would preclude protocol treatment
* No history of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that would contraindicate use of an investigational drug, affect the interpretation of the results of the study, or render the patient at high risk for treatment complications
* No clinically significant cardiac disease, including any of the following:

  * Uncontrolled hypertension (i.e., blood pressure > 150/100 mm Hg despite antihypertensive medication)
  * Myocardial infarction within the past year
  * Unstable angina
  * New York Heart Association class II-IV congestive heart failure
  * Unstable symptomatic arrhythmia requiring medication

    * Chronic atrial arrhythmia (i.e., atrial fibrillation or paroxysmal supraventricular tachycardia) allowed
* No clinically significant peripheral vascular disease
* No evidence of bleeding diathesis or coagulopathy
* No significant traumatic injury within the past 28 days
* No serious, nonhealing wound or ulcer, or concurrent healing fracture
* No history of aneurysm, stroke, transient ischemic attack, or arteriovenous malformation
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior treatment for pancreatic cancer
* More than 5 years since prior chemotherapy for malignancies other than pancreatic cancer
* No prior radiotherapy to the target volume
* More than 28 days since prior major surgical procedure or open biopsy
* At least 28 days since prior surgical bypass
* More than 7 days since prior fine-needle aspiration or core biopsy
* No prior organ transplant
* At least 4 weeks since prior sorivudine or brivudine
* At least 30 days since prior cimetidine
* No concurrent major surgical procedure

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2005-10-10 (Actual); Primary Completion 2007-12-17 (Actual); Study Completion 2010-07-16 (Actual)

PRIMARY OUTCOMES:
Response rate | After 10 weeks of concurrent therapy
  Response will be measured by CT scans using Recist and defined as Complete Response, Partial Response, Stable disease/no response, Progressive Disease.

SECONDARY OUTCOMES:
Toxicity profile of bevacizumab and gemcitabine with radiation therapy | After every cycle of therapy (cycle = 3-4 weeks), then every 3 months for 2 years, then every 6 months for 3 years, then yearly up to 10 years or until disease progression.
  Toxicities will be measured using National Cancer Institute's Common Toxicity Criteria for adverse events version 3.0 (CTCAE v3.0). Adverse events (AE)are graded:
  Grade 1 Mild AE Grade 2 Moderate AE Grade 3 Severe AE Grade 4 Life-threatening or disabling AE Grade 5 Death related to AE

CONTACTS AND LOCATIONS:
Overall Officials: William Small, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Result] Small W Jr, Mulcahy M, Benson A, et al.: A phase II trial of weekly gemcitabine and bevacizumab in combination with abdominal radiation therapy in patients with localized pancreatic cancer. [Abstract] J Clin Oncol 25 (Suppl 18): A-15043, 637s, 2007.
- [Derived] Rezai P, Yaghmai V, Tochetto SM, Galizia MS, Miller FH, Mulcahy MF, Small W Jr. Change in the growth rate of localized pancreatic adenocarcinoma in response to gemcitabine, bevacizumab, and radiation therapy on MDCT. Int J Radiat Oncol Biol Phys. 2011 Oct 1;81(2):452-9. doi: 10.1016/j.ijrobp.2010.05.060. Epub 2011 May 11. PMID 21570199